CLINICAL TRIAL: NCT00002161
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Adefovir Dipivoxil When Added to Standard Antiretroviral Therapy for the Treatment of HIV-Infected Patients With CD4 Cell Counts >= 200/mm3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 232C; GS-96-408
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-05

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Adenine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — adefovir dipivoxil

INTERVENTIONS:
Drug: Adefovir dipivoxil

SUMMARY:
To evaluate the anti-HIV activity, safety, and tolerance of adefovir dipivoxil ( bis-POM PMEA ) in combination with standard antiretroviral therapy for 48 weeks.

DETAILED DESCRIPTION:
Patients are randomized to receive either adefovir dipivoxil or placebo daily for 24 weeks, after which all patients will receive open-label drug for an additional 24 weeks. Study drug is administered in combination with a current antiretroviral regimen for the entire 48 weeks. Patients are followed every 4 weeks during the first 24 weeks of study, then every 8 weeks during the last 24 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection with HIV RNA titer >= 2500 copies/ml (2.5 KEq/ml) plasma.
* CD4 count >= 200 cells/mm3.
* No new AIDS-defining event within the past 2 months.
* Life expectancy at least 1 year.
* Consent of parent or guardian if less than 18 years old.
* Tolerated antiretroviral therapy for the past 2 months.

NOTE:

* Kaposi's sarcoma is permitted provided patient has not received systemic therapy within the past month.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active, serious infections other than HIV that require parenteral antibiotic or antiviral therapy.
* Gastrointestinal malabsorption syndrome or chronic nausea or vomiting that would preclude oral medication.
* Malignancy other than Kaposi's sarcoma or basal cell carcinoma.

Concurrent Medication:

Excluded:

* Immunomodulating agents such as systemic corticosteroids, IL-2, or interferons.
* Isoniazid.
* Rifampin.
* Investigational agents (unless approved by sponsor).
* Systemic chemotherapeutic agents.

Prior Medication:

Excluded:

* Parenteral antibiotic or antiviral therapy for another active, serious infection within the past 2 weeks.
* Immunomodulating agents such as systemic corticosteroids, IL-2, or interferons within the past month.
* Systemic therapy for KS within the past month.

Required:

* Antiretroviral regimen other than study drug.

Required:

* Antiretroviral therapy for at least the past 2 months. Current alcohol or substance abuse that would interfere with compliance.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - East Bay AIDS Ctr, Berkeley, California
  - Kraus Med Partners, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - San Mateo County Med Ctr / San Mateo County AIDS Prog, San Mateo, California
  - Pacific Oaks Research, Sherman Oaks, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Institute for Clinical Research, Washington D.C., District of Columbia
  - Univ of South Florida, St. Petersburg, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Northwestern Univ Med Ctr, Chicago, Illinois
  - Tulane Univ / Tulane / LSU Clinical Trials Unit, New Orleans, Louisiana
  - Harvard Univ / Massachusetts Gen Hosp, Boston, Massachusetts
  - Wayne State Univ / Univ Health Ctr, Detroit, Michigan
  - Albany Med College / Clinical Pharmacy Studies, Albany, New York
  - Saint Vincent's Med Ctr, New York, New York
  - Carolinas Med Ctr, Charlotte, North Carolina
  - The Research and Education Group, Portland, Oregon
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Dallas VA Med Ctr, Dallas, Texas
  - Univ of Texas, Galveston, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Univ of Utah School of Medicine, Salt Lake City, Utah
  - Univ of Wisconsin, Madison, Wisconsin